CLINICAL TRIAL: NCT00280540
Title: A 6-week Treatment Regimen Study to Evaluate the Efficacy of Initial High Dose Valsartan Monotherapy (160 mg) or Combo Therapy (Valsartan + Hydrochlorothiazide, 160/12.5 mg) to Conventional Low-dose Valsartan Monotherapy (80 mg) in Managing Patients With Hypertension
Brief Title: Efficacy and Safety of Valsartan/Hydrochlorothiazide Combination Therapy in Patients With Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CVAH631BUS05
Record Dates: First submitted 2006-01-19; First posted 2006-01-23 (Estimated); Last update posted 2010-11-09 (Estimated); Status verified 2008-03

CONDITIONS: Hypertension
Keywords: Hypertension; High blood pressure; Blood pressure control; Blood pressure reduction; Valsartan
MeSH Terms: conditions — Hypertension | interventions — Valsartan; Hydrochlorothiazide

INTERVENTIONS:
Drug: Valsartan/Hydrochlorothiazide

SUMMARY:
This is a double-blind study to evaluate the reduction in systolic blood pressure using a therapy initiated with valsartan 160 mg or valsartan + hydrochlorothiazide (HCTZ) 160/12.5 mg compared to a more conventional approach (therapy initiated with low-dose valsartan 80 mg).

ELIGIBILITY:
Inclusion Criteria:

* Male or female age 18 or older
* Diagnosed as having hypertension (mean seated systolic blood pressure ≥ 150 mm Hg but < 180 mm Hg and mean seated diastolic blood pressure ≥ 90 mm Hg and <110 mm Hg)

Exclusion Criteria:

* Patients with severe hypertension: Systolic ≥ 180 mm Hg or Diastolic ≥ 110 mm Hg
* History of secondary hypertension (including primary aldosteronism, renovascular hypertension, pheochromocytoma etc.)
* History of myocardial infarction, stroke [e.g. cerebrovascular accident (CVA), thrombotic stroke, transient ischemic attack (TIA)], or onset of heart failure within the last 6 months.

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 648
Dates: Start 2005-12; Primary Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline systolic blood pressure after 4 weeks
Change from baseline systolic blood pressure after 2 and 6 weeks

SECONDARY OUTCOMES:
Time in weeks to achieve blood pressure less than 140/90 mmHg over 6 week period
Blood pressure less than 140/90 mmHg after 6 weeks
Change from baseline diastolic blood pressure after 6 weeks
Change from baseline in blood and urine markers after 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis
Locations (1):
- Novartis Pharmaceuticals, East Hanover, New Jersey, United States

REFERENCES:
- [Derived] Zappe DH, Palmer BF, Calhoun DA, Purkayastha D, Samuel R, Jamerson KA. Effectiveness of initiating treatment with valsartan/hydrochlorothiazide in patients with stage-1 or stage-2 hypertension. J Hum Hypertens. 2010 Jul;24(7):483-91. doi: 10.1038/jhh.2009.90. Epub 2009 Dec 10. PMID 20010618